CLINICAL TRIAL: NCT03365934
Title: Randomized, Exploratory Study to Evaluate Changes to Skin Microbiome With Tape-stripped Wounds
Brief Title: Evaluation of Changes to Skin Microbiome With Tape-Stripped Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-170726100607-SACT
Record Dates: First submitted 2017-11-16; First posted 2017-12-08 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Microflora; Microbiome; skin physiology; Fitzpatrick Skin Types I-III; Tape-stripped wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- ADHESIVE BANDAGE #1 (Experimental): bandage applied to wounded site.
  Interventions: Device: ADHESIVE BANDAGE #1
- ADHESIVE BANDAGE #2 (Experimental): bandage applied to wounded site.
  Interventions: Device: ADHESIVE BANDAGE #2
- ADHESIVE BANDAGE #3 (Experimental): bandage applied to wounded site
  Interventions: Device: ADHESIVE BANDAGE #3
- Antibacterial Bandage with 0.8% BZK (Experimental): bandage with 0.8% Benzalkonium Chloride (BZK) applied to wounded site
  Interventions: Device: Antibacterial Bandage with 0.8% BZK
- Intact and No Bandage (Other): This test site will remain intact (not wounded) and not treated with a bandage, serving as a negative control site.
  Interventions: Other: Intact and No Bandage
- Wounded and No Bandage (Other): This test site will be wounded and no bandage applied, serving as a positive control site.
  Interventions: Other: Wounded and No Bandage

INTERVENTIONS:
Device: ADHESIVE BANDAGE #1 — Bandage applied daily to wounded site for 14 days
  Arms: ADHESIVE BANDAGE #1
Device: ADHESIVE BANDAGE #2 — Bandage applied daily to wounded site for 14 days
  Arms: ADHESIVE BANDAGE #2
Device: ADHESIVE BANDAGE #3 — Bandage applied daily to wounded site for 14 days
  Arms: ADHESIVE BANDAGE #3
Device: Antibacterial Bandage with 0.8% BZK — bandage with 0.8% Benzalkonium Chloride (BZK) applied daily to wounded site for 14 days
  Arms: Antibacterial Bandage with 0.8% BZK
Other: Intact and No Bandage — This test site will remain intact (not wounded) and not treated with a bandage, serving as a negative control site.
  Arms: Intact and No Bandage
Other: Wounded and No Bandage — This test site will be wounded but will not be treated with a bandage, serving as the positive control site.
  Arms: Wounded and No Bandage

SUMMARY:
This single center, randomized, 15-day clinical trial is being conducted to assess the changes to the skin microbiome of induced wounds on the back in approximately 35 healthy adult subjects aged 18-55 years, with Fitzpatrick Skin Types I - III. Microbiome and skin physiology assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 55 years of age.
2. Fitzpatrick skin types I to III.
3. Must be able to comprehend and follow the requirements of the study
4. Avoid excessive sun exposure
5. Willing to refrain from topical product use on the back for the duration of the study.
6. Subjects must agree not to immerse their bandages in water for the duration of the study.
7. Male and female subjects with reproductive potential who agree to practice a medically acceptable form of birth control

Exclusion Criteria:

1. Excessively hairy back, acne, scars and pigmentation or nevi t
2. . Pregnant or Lactating, or planning on becoming pregnant;
3. . Known allergies or sensitivities to anesthetics, adhesive bandages, wound treatment products or tapes;
4. . Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results
5. Participation in any other clinical study within 30 days of Visit 1;
6. . Subjects who have a health condition and/or pre-existing or dormant dermatologic conditions or who have clinically active bacterial, fungal, or viral skin infections or those who are susceptible to cutaneous infections
7. Subjects who report using prescription or OTC medication (oral or topical) that can make skin more sensitive or influence the skin (i.e. antibiotics, hormones, insulin, etc.)
8. Subjects receiving topical and/or inhaled medications that may alter or compromise the bleeding/healing process
9. Individuals with a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications and/or radiation
10. . Subjects with a known history of keloid or hypertrophic scar formation;
11. Subjects diagnosed with any blood clotting disorder;
12. Hyperthyroidism or hypothyroidism or with active or recently treated (within 1 year) skin cancer, or those in poor nutritional status; 13 Subjects taking oral Vitamin A derivatives such as Accutane, isotretinon, or using retinoic acid in the past 1 year or using topical Vitamin A derivatives in the 3 weeks prior to study start;

14. Subjects with clinically infected skin lesions; 15. Subjects with cracked or excoriated skin, or other skin problems. 16. Diabetes mellitus that cannot be controlled by diet alone (i.e. requires systemic medications for control); 17. Subjects with friable skin, at the discretion of the Investigator;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lastella, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research Inc., Fair Lawn, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Randomized Subjects: All Randomized Subjects
Period: Overall Study
Arm/Group | All Randomized Subjects
Started | 35
Completed | 33
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America: USA | 35

OUTCOME MEASURES:

1. Primary Outcome: Microbial Community Richness - Baseline (Day 0)
Description: Swabs will be collected on the back at Baseline (Day 0) and analyzed to determine the total number of different bacterial taxa (microorganisms) detected in the sample. There was no prespecified primary endpoint in the protocol.
Time Frame: Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Groups:
- Intact Uncovered Skin: Intact Uncovered Skin
- Wounded Uncovered Skin: Wounded Uncovered Skin
- Product #1: Product #1
- Product #2: Product #2
- Product #3: Product #3
- Product #4: Product #4
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 22 | 28 | 27 | 23 | 27
Number of bacterial taxa | 56.5862069 [41.82700101 to 71.34541279] | 32.13043478 [21.71828318 to 42.54258639] | 43.72413793 [31.41567266 to 56.0326032] | 34.03703704 [25.21769482 to 42.85637925] | 42.39130435 [28.2925728 to 56.4900359] | 46.48148148 [32.28761284 to 60.67535013]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.071225, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.092027, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.601716, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.639911, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.842476, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.999941, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.883479, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.782208, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.607134, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.939549, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.86475, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.704759, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.999989, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.997568, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999518, t-test, 2 sided

2. Primary Outcome: Microbial Community Richness - (Day 1)
Description: Swabs will be collected on the back at Day 1 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 29 | 27 | 32 | 19 | 24
Number of bacterial taxa | 53.15625 [38.21010189 to 68.10239811] | 58.75862069 [47.10408916 to 70.41315222] | 22 [18.01079945 to 25.98920055] | 53.5 [37.61649637 to 69.38350363] | 42.47368421 [27.00391618 to 57.94345224] | 28.83333333 [20.99591479 to 36.67075187]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.985332, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.870459, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.004963, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.071935, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.988995, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.545378, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000649, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.014600, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.854566, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.004322, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.0651, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.300536, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.753883, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.97621, t-test, 2 sided

3. Primary Outcome: Microbial Community Richness - (Day 2)
Description: Swabs will be collected on the back at Day 2 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 33 | 33 | 32 | 27 | 32
Number of bacterial taxa | 60.15625 [45.95442154 to 74.35807846] | 87.03030303 [64.50676969 to 109.5538364] | 20.33333333 [15.69936368 to 24.96730299] | 36.65625 [30.26643624 to 43.04606376] | 33.7037037 [22.14710131 to 45.2603061] | 30.40625 [23.74762413 to 37.06487587]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.027774, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.08431, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.049247, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000126, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.010829, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999533, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.4205363, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.9802252, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.6845362, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.9992002, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.8562779, t-test, 2 sided

4. Primary Outcome: Microbial Community Richness - (Day 3)
Description: Swabs will be collected on the back at Day 3 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 32 | 33 | 27 | 25 | 32
Number of bacterial taxa | 53.44827586 [40.61259145 to 66.28396027] | 74.03125 [60.80846371 to 87.25403629] | 19.21212121 [16.49174219 to 21.93250024] | 38.25925926 [29.78367344 to 46.73484508] | 37.88 [23.44927006 to 52.31072994] | 30.28125 [23.87137083 to 36.69112917]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.0403539, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.2953049, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.290551, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.0000247, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.0133001, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.0000167, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.0000212, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.99999995, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.0792013, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.870163, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.103828, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.900265, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.570015, t-test, 2 sided

5. Primary Outcome: Microbial Community Richness - (Day 4)
Description: Swabs will be collected on the back at Day 4 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 4
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 26 | 30 | 32 | 31 | 28 | 32
Number of bacterial taxa | 66.88461538 [47.31497155 to 86.45425922] | 76.23333333 [61.4245631 to 91.04210357] | 20.5 [17.18168127 to 23.81831873] | 44.35483871 [33.45042213 to 55.25925529] | 43.53571429 [29.33570468 to 57.73572389] | 25.59375 [20.71187082 to 30.47562918]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.882449, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.088558, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.081846, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.0000303, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.001817, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.001825, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999999, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.038836, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.184508, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.062829, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.253458, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.987798, t-test, 2 sided

6. Primary Outcome: Microbial Community Richness - (Day 5)
Description: Swabs will be collected on the back at Day 5 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 5
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 25 | 27 | 31 | 27 | 21 | 31
Number of bacterial taxa | 61.96 [44.36091054 to 79.55908946] | 77.59259259 [60.00060441 to 95.18458078] | 19.03225806 [16.42738215 to 21.63713398] | 44.03703704 [29.83167678 to 58.2423973] | 50.33333333 [32.41789542 to 68.24877125] | 25.80645161 [21.1508763 to 30.46202693]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.516068, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.358412, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.834145, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000035, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000843, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.002997, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.051717, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.985602, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.046422, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.28061, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.011015, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.089156, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.963882, t-test, 2 sided

7. Primary Outcome: Microbial Community Richness - (Day 6)
Description: Swabs will be collected on the back at Day 6 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 6
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 18 | 27 | 29 | 27 | 19 | 30
Number of bacterial taxa | 48.5 [35.54549519 to 61.45450481] | 75.88888889 [61.54822817 to 90.2295496] | 23.55172414 [20.03657535 to 27.06687293] | 48.81481481 [37.40801959 to 60.22161004] | 40.26315789 [26.53167948 to 53.99463631] | 25.63333333 [21.01769583 to 30.24897084]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.00526, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.914409, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.013004, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.028517, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.001356, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.000059, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.859272, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.002821, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.007492, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.208803, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.341884, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999531, t-test, 2 sided

8. Primary Outcome: Microbial Community Richness - (Day 7)
Description: Swabs will be collected on the back at Day 7 and analyzed to determine the total number of different bacteria Taxa (microorganismss) detected in the sample.
Time Frame: Day 7
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 22 | 33 | 31 | 25 | 21 | 33
Number of bacterial taxa | 54.54545455 [40.08770259 to 69.0032065] | 81.51515152 [62.74620188 to 100.2841011] | 31 [23.08861196 to 38.91138804] | 45.12 [28.23285287 to 62.00714713] | 43.04761905 [27.89745068 to 58.19778741] | 30.57575758 [24.32822886 to 36.82328629]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.066788, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.942653, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.893545, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.165225, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.140475, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.002026, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.001916, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999957, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.672573, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.630145, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.832757, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.803277, t-test, 1 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 1, t-test, 2 sided

9. Primary Outcome: Microbial Community Richness - (Day 14)
Description: Swabs will be collected on the back at Day 14 and analyzed to determine the total number of different bacteria Taxa (microorganisms) detected in the sample.
Time Frame: Day 14
Measure: Mean (95% Confidence Interval); unit: Number of bacterial taxa
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 30 | 27 | 32 | 32 | 25 | 33
Number of bacterial taxa | 73.1 [57.23395854 to 88.96604146] | 66.44444444 [48.7698287 to 84.11906019] | 28.34375 [24.26615289 to 32.42134711] | 46.21875 [39.38246899 to 53.05503101] | 32.32 [25.7083049 to 38.9316951] | 30.45454545 [25.6128987 to 35.29619221]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.943522, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.002376, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.061015, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.000211, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.412626, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.104388, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.197791, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.994413, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.999851, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999621, t-test, 2 sided

10. Primary Outcome: Microbial Community Diversity - Baseline (Day 0)
Description: Swabs will be collected on the back at Baseline (Day 0) for analysis based on the Shannon Index.
Time Frame: Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 22 | 28 | 27 | 23 | 27
Shannon Diversity Index | 1.702946961 [1.212183074 to 2.193710849] | 0.938913363 [0.465348751 to 1.412477975] | 1.470084856 [1.011374271 to 1.928795441] | 1.16250018 [0.709007612 to 1.615992753] | 1.355575793 [0.832569386 to 1.8785822] | 1.278886018 [0.840487425 to 1.717284611]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.193667, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.526573, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.898749, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.975044, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.760706, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.985237, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.837995, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.592697, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.912495, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.99245, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.925553, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.999171, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.999324, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.999913, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.990516, t-test, 2 sided

11. Primary Outcome: Microbial Community Diversity - Day 1
Description: Swabs will be collected on the back at Day 1 for analysis based on the Shannon Index.
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 29 | 27 | 32 | 19 | 24
Shannon Diversity Index | 1.703357647 [1.261265404 to 2.145449891] | 1.45014401 [1.047686471 to 1.852601549] | 0.786918525 [0.546103958 to 1.027733092] | 1.518890457 [1.116626746 to 1.921154169] | 1.060560749 [0.544639084 to 1.576482413] | 0.900390717 [0.622715277 to 1.178066157]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.92106, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.976812, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.233992, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.007591, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.038958, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.99809, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.773028, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.135805, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.350556, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.61046, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.062163, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.203418, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.942304, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.995238, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.99858, t-test, 2 sided

12. Primary Outcome: Microbial Community Diversity - Day 2
Description: Swabs will be collected on the back at Day 2 for analysis based on the Shannon Index.
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 33 | 33 | 32 | 27 | 32
Shannon Diversity Index | 1.776794637 [1.324060973 to 2.229528302] | 1.866171013 [1.449444421 to 2.282897605] | 0.793586986 [0.62136427 to 0.965809702] | 1.169519236 [0.888383719 to 1.450654753] | 1.327096148 [0.903682194 to 1.750510103] | 0.941432164 [0.692964696 to 1.189899633]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.998949, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.111084, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.456846, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.00062, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.006871, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.039407, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.245375, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000113, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.001612, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.988067, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.599171, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.928722, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.256079, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.626498, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.988693, t-test, 2 sided

13. Primary Outcome: Microbial Community Diversity - Day 3
Description: Swabs will be collected on the back at Day 3 for analysis based on the Shannon Index.
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 32 | 33 | 27 | 25 | 32
Shannon Diversity Index | 1.85115546 [1.382317602 to 2.319993318] | 1.765408531 [1.338653068 to 2.192163994] | 0.7122095 [0.538547591 to 0.885871409] | 1.046670711 [0.736643325 to 1.356698098] | 1.322070974 [0.943427192 to 1.700714756] | 1.071628134 [0.813088017 to 1.330168251]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.99916, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.016246, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.289112, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000038, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.014558, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.03731, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.465745, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000112, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.034575, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.889597, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.726932, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.999998, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.130235, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.910989, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.616933, t-test, 2 sided

14. Primary Outcome: Microbial Community Diversity - Day 4
Description: Swabs will be collected on the back at Day 4 for analysis based on the Shannon Index.
Time Frame: Day 4
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 26 | 30 | 32 | 31 | 28 | 32
Shannon Diversity Index | 1.932633093 [1.431535105 to 2.433731082] | 1.88044173 [1.433470325 to 2.327413134] | 0.797557627 [0.628526357 to 0.966588896] | 1.453888326 [1.117071932 to 1.790704721] | 1.513528952 [1.052864028 to 1.974193877] | 0.76492761 [0.567335326 to 0.962519895]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.999952, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.421347, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.598141, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000197, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000115, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.511155, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.693868, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000232, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000133, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999894, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.078046, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.054975, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.050132, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.034793, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999993, t-test, 2 sided

15. Primary Outcome: Microbial Community Diversity - Day 5
Description: Swabs will be collected on the back at Day 5 for analysis based on the Shannon Index.
Time Frame: Day 5
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 25 | 27 | 31 | 27 | 21 | 31
Shannon Diversity Index | 1.783329786 [1.22306299 to 2.343596582] | 1.664197367 [1.212563987 to 2.115830748] | 0.700642641 [0.529568098 to 0.871717184] | 1.267584901 [0.901217742 to 1.633952061] | 1.480613855 [0.994345968 to 1.966881743] | 0.68710958 [0.515014462 to 0.859204698]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.997406, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.354187, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.883222, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000412, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000332, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.626878, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.984465, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.001845, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.001507, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.970029, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.19886, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.177549, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.041698, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.036131, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 1, t-test, 2 sided

16. Primary Outcome: Microbial Community Diversity - Day 6
Description: Swabs will be collected on the back at Day 6 for analysis based on the Shannon Index.
Time Frame: Day 6
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 18 | 27 | 29 | 27 | 19 | 30
Shannon Diversity Index | 1.782776526 [1.184618285 to 2.380934768] | 1.799754753 [1.346147213 to 2.253362293] | 0.865721173 [0.642359805 to 1.089082541] | 1.223240388 [0.927644983 to 1.518835794] | 1.425318411 [0.881697663 to 1.968939159] | 0.698409234 [0.484505139 to 0.912313329]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.317315, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.829352, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.010561, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.001099, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.175148, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.728796, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.001992, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000113, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.974567, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.668933, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.239446, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.283848, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.06829, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.979516, t-test, 2 sided

17. Primary Outcome: Microbial Community Diversity - Day 7
Description: Swabs will be collected on the back at Day 7 for analysis based on the Shannon Index.
Time Frame: Day 7
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 22 | 33 | 31 | 25 | 21 | 33
Shannon Diversity Index | 1.637800497 [1.118090334 to 2.15751066] | 1.765588383 [1.340278816 to 2.190897951] | 0.848189016 [0.629210776 to 1.067167257] | 1.328769036 [0.915319287 to 1.742218786] | 1.367835908 [0.901653933 to 1.834017883] | 0.791935871 [0.565396501 to 1.018475241]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.996522, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.875832, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.938, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.038527, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.018334, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.512209, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.665529, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.002257, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000728, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999993, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.417914, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.277469, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.385419, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.257647, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999897, t-test, 2 sided

18. Primary Outcome: Microbial Community Diversity - Day 14
Description: Swabs will be collected on the back at Day 14 for analysis based on the Shannon Index.
Time Frame: Day 14
Measure: Mean (95% Confidence Interval); unit: Shannon Diversity Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 30 | 27 | 32 | 32 | 25 | 33
Shannon Diversity Index | 1.992920174 [1.528772641 to 2.457067706] | 1.729295419 [1.273786002 to 2.184804836] | 0.826824832 [0.642994336 to 1.010655328] | 1.188271444 [0.950876818 to 1.42566607] | 1.362870394 [0.978315938 to 1.747424849] | 0.729090928 [0.540015069 to 0.918166787]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.862516, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.00473, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.085238, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.168409, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.652654, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.001436, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000235, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.974842, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.557877, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.277244, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.195527, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.070843, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.997565, t-test, 2 sided

19. Primary Outcome: Microbial Community Evenness - Baseline (Day 0)
Description: Swabs will be collected on the back at Baseline (Day 0) for analysis based on the Pielou's Evenness Index.
Time Frame: Day 0
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 22 | 28 | 27 | 23 | 27
Pielou's Evenness Index | 0.410155753 [0.305407316 to 0.51490419] | 0.271955307 [0.143543228 to 0.400367386] | 0.402950073 [0.37196059 to 0.518890538] | 0.320061269 [0.201925423 to 0.438197114] | 0.358334602 [0.228095257 to 0.488573947] | 0.325047059 [0.217282735 to 0.432811384]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.016628, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.217862, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.812915, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.999971, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.275557, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.870124, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.380144, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.029518, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.815476, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.944307, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.313389, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.999996, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.894272, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.969093, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.383434, t-test, 2 sided

20. Primary Outcome: Microbial Community Evenness - Day 1
Description: Swabs will be collected on the back at Day 1 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 29 | 27 | 32 | 19 | 24
Pielou's Evenness Index | 0.437132278 [0.330359027 to 0.54390553] | 0.349459879 [0.255994131 to 0.442925627] | 0.246062404 [0.173290416 to 0.318834392] | 0.389333736 [0.294031092 to 0.484636381] | 0.273028286 [0.154944552 to 0.391112019] | 0.265726584 [0.192716814 to 0.338736354]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.393119, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.890335, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.021978, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000983, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.006615, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.951883, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.692455, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.257254, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.530181, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.219274, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.029675, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.111454, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.995849, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.999994, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.998744, t-test, 2 sided

21. Primary Outcome: Microbial Community Evenness - Day 2
Description: Swabs will be collected on the back at Day 2 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 33 | 33 | 32 | 27 | 32
Pielou's Evenness Index | 0.42693493 [0.32874755 to 0.52512231] | 0.415386732 [0.332645201 to 0.498128264] | 0.263575452 [0.212813889 to 0.314337015] | 0.322568391 [0.249971799 to 0.395164982] | 0.386309873 [0.276870199 to 0.495749548] | 0.277342605 [0.212258941 to 0.342426269]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.999858, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.215132, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.958812, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.00622, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.017733, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.330576, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.990334, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.013025, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.034707, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.771698, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.790117, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.923224, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.112245, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.216229, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999663, t-test, 2 sided

22. Primary Outcome: Microbial Community Evenness - Day 3
Description: Swabs will be collected on the back at Day 3 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 32 | 33 | 27 | 25 | 32
Pielou's Evenness Index | 0.455666826 [0.348282864 to 0.563050789] | 0.405262792 [0.310526103 to 0.49999948] | 0.234966957 [0.183226948 to 0.286706967] | 0.279414327 [0.204200672 to 0.354627983] | 0.363143499 [0.268134344 to 0.458152655] | 0.312661752 [0.250785086 to 0.374538417]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.91874, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.013582, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.523284, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000315, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.059485, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.15037, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.967277, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.008729, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.421603, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.647267, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.953645, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.987387, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.147361, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.930371, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.6094, t-test, 2 sided

23. Primary Outcome: Microbial Community Evenness - Day 4
Description: Swabs will be collected on the back at Day 4 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 4
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 26 | 30 | 32 | 31 | 28 | 32
Pielou's Evenness Index | 0.451377803 [0.350796707 to 0.5519589] | 0.422737764 [0.328361231 to 0.517114298] | 0.269049335 [0.216107994 to 0.321990676] | 0.38804873 [0.312100017 to 0.463997444] | 0.392633921 [0.288519448 to 0.496748395] | 0.231556861 [0.177760893 to 0.285352829]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.99253, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.795279, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.855067, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.003915, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000221, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.97816, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.98972, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.01764, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.001185, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999999, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.119961, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.013468, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.112192, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.013135, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.965966, t-test, 2 sided

24. Primary Outcome: Microbial Community Evenness - Day 5
Description: Swabs will be collected on the back at Day 5 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 5
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 25 | 27 | 31 | 27 | 21 | 31
Pielou's Evenness Index | 0.418779366 [0.300422474 to 0.537136258] | 0.377673266 [0.28316356 to 0.472182971] | 0.235666776 [0.181164664 to 0.290168889] | 0.330181203 [0.249683185 to 0.410679222] | 0.388971323 [0.268970894 to 0.508971751] | 0.212340111 [0.163649748 to 0.261030475]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.968005, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.526293, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.994384, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.004967, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000948, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.936394, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.999945, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.050032, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.01256, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.886978, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.391295, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.163678, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.047937, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.013231, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.996358, t-test, 2 sided

25. Primary Outcome: Microbial Community Evenness - Day 6
Description: Swabs will be collected on the back at Day 6 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 6
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 18 | 27 | 29 | 27 | 19 | 30
Pielou's Evenness Index | 0.446298915 [0.307295525 to 0.585302305] | 0.417003638 [0.315872307 to 0.51813497] | 0.270297461 [0.208318912 to 0.33227601] | 0.31595456 [0.242353894 to 0.389555227] | 0.370960196 [0.242456263 to 0.499464128] | 0.213078749 [0.150385636 to 0.275771862]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.995862, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.223341, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.834338, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.030267, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.00104, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.377217, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.965547, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.052284, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.001348, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.927936, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.946487, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.327918, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.475038, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.060057, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.857177, t-test, 2 sided

26. Primary Outcome: Microbial Community Evenness - Day 7
Description: Swabs will be collected on the back at Day 7 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 7
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 22 | 33 | 31 | 25 | 21 | 33
Pielou's Evenness Index | 0.410567291 [0.286544213 to 0.534590369] | 0.404030653 [0.309872763 to 0.498188542] | 0.247507869 [0.190648545 to 0.304367193] | 0.354717133 [0.259034665 to 0.450399602] | 0.359914043 [0.242240002 to 0.477588085] | 0.230659131 [0.174438405 to 0.286879856]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.999997, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.938793, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.965993, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.057803, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.022816, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.945179, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.972522, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.033704, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.010747, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.999999, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.385474, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.213798, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.388682, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.22386, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.999494, t-test, 2 sided

27. Primary Outcome: Microbial Community Evenness - Day 14
Description: Swabs will be collected on the back at Day 14 for analysis based on the Pielou's Evenness Index.
Time Frame: Day 14
Measure: Mean (95% Confidence Interval); unit: Pielou's Evenness Index
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 30 | 27 | 32 | 32 | 25 | 33
Pielou's Evenness Index | 0.454253238 [0.360645958 to 0.547860518] | 0.402829439 [0.309226175 to 0.496432702] | 0.249502521 [0.196421318 to 0.302583723] | 0.308795465 [0.25494207 to 0.362648861] | 0.383110745 [0.283994153 to 0.482227337] | 0.210741952 [0.159426533 to 0.262057372]
Statistical Analysis 1: Comparison: Intact Uncovered Skin vs Wounded Uncovered Skin; Test type: Superiority; p = 0.891244, t-test, 2 sided
Statistical Analysis 2: Comparison: Intact Uncovered Skin vs Product #2; Test type: Superiority; p = 0.022659, t-test, 2 sided
Statistical Analysis 3: Comparison: Intact Uncovered Skin vs Product #3; Test type: Superiority; p = 0.693615, t-test, 2 sided
Statistical Analysis 4: Comparison: Intact Uncovered Skin vs Product #1; Test type: Superiority; p = 0.000237, t-test, 2 sided
Statistical Analysis 5: Comparison: Intact Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000005, t-test, 2 sided
Statistical Analysis 6: Comparison: Wounded Uncovered Skin vs Product #2; Test type: Superiority; p = 0.352008, t-test, 2 sided
Statistical Analysis 7: Comparison: Wounded Uncovered Skin vs Product #3; Test type: Superiority; p = 0.998761, t-test, 2 sided
Statistical Analysis 8: Comparison: Wounded Uncovered Skin vs Product #1; Test type: Superiority; p = 0.017832, t-test, 2 sided
Statistical Analysis 9: Comparison: Wounded Uncovered Skin vs Product #4; Test type: Superiority; p = 0.000974, t-test, 2 sided
Statistical Analysis 10: Comparison: Product #2 vs Product #3; Test type: Superiority; p = 0.638238, t-test, 2 sided
Statistical Analysis 11: Comparison: Product #1 vs Product #2; Test type: Superiority; p = 0.777423, t-test, 2 sided
Statistical Analysis 12: Comparison: Product #2 vs Product #4; Test type: Superiority; p = 0.249909, t-test, 2 sided
Statistical Analysis 13: Comparison: Product #1 vs Product #3; Test type: Superiority; p = 0.068196, t-test, 2 sided
Statistical Analysis 14: Comparison: Product #3 vs Product #4; Test type: Superiority; p = 0.005786, t-test, 2 sided
Statistical Analysis 15: Comparison: Product #1 vs Product #4; Test type: Superiority; p = 0.954163, t-test, 2 sided

28. Secondary Outcome: Skin Barrier Function -Baseline (Day 0)
Description: The skin barrier function of the test sites will be evaluated at Baseline (Day 0) by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
g/m^2/hr | 9.82 (6.725) | 96.94 (11.682) | 101.08 (9.992) | 97.04 (13.397) | 101.43 (11.116) | 98.21 (13.165)

29. Secondary Outcome: Skin Barrier Function - Day 1
Description: The skin barrier function of the test sites will be evaluated at Day 1 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34
g/m^2/hr | 13.05 (13.414) | 95.68 (16.393) | 92.40 (10.886) | 91.13 (14.689) | 97.91 (14.527) | 97.61 (15.420)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 1; Test type: Superiority; p = 0.009, ANCOVA; Mean Difference (Net) = -7.50, 95% CI 2-sided [-13.1279 to -1.8688], Standard Error of Mean 2.851
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 1; Test type: Superiority; p = 0.077, ANCOVA; Mean Difference (Net) = -5.08, 95% CI 2-sided [-10.7083 to 0.5508], Standard Error of Mean 2.851
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 1; Test type: Superiority; p = 0.399, ANCOVA; Mean Difference (Net) = -2.41, 95% CI 2-sided [-8.0399 to 3.2192], Standard Error of Mean 2.851
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 1; Test type: Superiority; p = 0.802, ANCOVA; Mean Difference (Net) = 0.72, 95% CI 2-sided [-4.9144 to 6.3446], Standard Error of Mean 2.851

30. Secondary Outcome: Skin Barrier Function - Day 2
Description: The skin barrier function of the test sites will be evaluated at Day 2 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33
g/m^2/hr | 10.97 (7.527) | 80.26 (22.229) | 73.10 (16.557) | 68.36 (20.387) | 82.63 (17.149) | 89.77 (17.470)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.37, 95% CI 2-sided [-17.3738 to -5.3723], Standard Error of Mean 3.038
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -12.68, 95% CI 2-sided [-18.6789 to -6.6775], Standard Error of Mean 3.038
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 2; Test type: Superiority; p = 0.521, ANCOVA; Mean Difference (Net) = -1.96, 95% CI 2-sided [-7.9571 to 4.0444], Standard Error of Mean 3.038
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 2; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Net) = 8.39, 95% CI 2-sided [2.3925 to 14.3940], Standard Error of Mean 3.038

31. Secondary Outcome: Skin Barrier Function - Day 3
Description: The skin barrier function of the test sites will be evaluated at Day 3 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33
g/m^2/hr | 15.46 (18.864) | 77.40 (24.567) | 50.41 (23.291) | 50.81 (20.377) | 68.49 (27.025) | 89.27 (18.969)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 3; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -31.83, 95% CI 2-sided [-41.3967 to -22.2538], Standard Error of Mean 4.847
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 3; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -27.30, 95% CI 2-sided [-36.8727 to -17.7298], Standard Error of Mean 4.847
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 3; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Net) = -13.71, 95% CI 2-sided [-23.2784 to -4.1355], Standard Error of Mean 4.847
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 3; Test type: Superiority; p = 0.039, ANCOVA; Mean Difference (Net) = 10.07, 95% CI 2-sided [0.4969 to 19.6398], Standard Error of Mean 4.847

32. Secondary Outcome: Skin Barrier Function - Day 4
Description: The skin barrier function of the test sites will be evaluated at Day 4 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34
g/m^2/hr | 16.70 (19.227) | 72.49 (25.078) | 36.32 (35.19) | 35.19 (20.969) | 56.14 (28.921) | 82.46 (28.101)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -40.39, 95% CI 2-sided [-51.0324 to -29.7496], Standard Error of Mean 5.390
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -37.84, 95% CI 2-sided [-48.4787 to -27.1959], Standard Error of Mean 5.390
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -20.99, 95% CI 2-sided [-31.6336 to -10.3508], Standard Error of Mean 5.390
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 4; Test type: Superiority; p = 0.106, ANCOVA; Mean Difference (Net) = 8.75, 95% CI 2-sided [-1.8871 to 19.3957], Standard Error of Mean 5.390

33. Secondary Outcome: Skin Barrier Function - Day 5
Description: The skin barrier function of the test sites will be evaluated at Day 5 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33
g/m^2/hr | 12.77 (16.829) | 58.87 (25.914) | 30.80 (21.510) | 32.27 (23.068) | 44.91 (32.510) | 67.46 (27.159)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 5; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -32.90, 95% CI 2-sided [-43.3249 to -22.4838], Standard Error of Mean 5.276
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 5; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -27.31, 95% CI 2-sided [-37.7279 to -16.8868], Standard Error of Mean 5.276
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 5; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -18.76, 95% CI 2-sided [-29.1785 to -8.3374], Standard Error of Mean 5.276
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 5; Test type: Superiority; p = 0.200, ANCOVA; Mean Difference (Net) = 6.79, 95% CI 2-sided [-3.6303 to 17.2107], Standard Error of Mean 5.276

34. Secondary Outcome: Skin Barrier Function - Day 6
Description: The skin barrier function of the test sites will be evaluated at Day 6 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 6
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
g/m^2/hr | 11.94 (8.699) | 47.34 (20.318) | 21.28 (8.524) | 22.81 (11.897) | 31.57 (17.810) | 53.56 (28.390)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 6; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -30.90, 95% CI 2-sided [-39.5325 to -22.2650], Standard Error of Mean 4.371
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 6; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -25.33, 95% CI 2-sided [-33.9669 to -16.6993], Standard Error of Mean 4.371
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 6; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -20.63, 95% CI 2-sided [-29.2588 to -11.9912], Standard Error of Mean 4.371
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 6; Test type: Superiority; p = 0.330, ANCOVA; Mean Difference (Net) = 4.27, 95% CI 2-sided [-4.3620 to 12.9055], Standard Error of Mean 4.371

35. Secondary Outcome: Skin Barrier Function - Day 7
Description: The skin barrier function of the test sites will be evaluated at Day 7 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33
g/m^2/hr | 9.80 (4.252) | 30.36 (16.556) | 21.23 (12.719) | 19.52 (7.545) | 25.08 (17.171) | 39.03 (25.197)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 7; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -13.95, 95% CI 2-sided [-21.3680 to -6.5419], Standard Error of Mean 3.754
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 7; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -11.54, 95% CI 2-sided [-18.9563 to -4.1302], Standard Error of Mean 3.754
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 7; Test type: Superiority; p = 0.008, ANCOVA; Mean Difference (Net) = -10.07, 95% CI 2-sided [-17.4867 to -2.6606], Standard Error of Mean 3.754
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 7; Test type: Superiority; p = 0.069, ANCOVA; Mean Difference (Net) = 6.87, 95% CI 2-sided [-0.5447 to 14.2814], Standard Error of Mean 3.754

36. Secondary Outcome: Skin Barrier Function - Day 14
Description: The skin barrier function of the test sites will be evaluated at Day 14 by Trans Epidermal Water Loss (TEWL).
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33
g/m^2/hr | 10.32 (14.697) | 14.58 (13.016) | 16.66 (9.356) | 16.10 (15.442) | 10.07 (4.165) | 16.45 (5.432)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #1 group based on the change from baseline at Day 14; Test type: Superiority; p = 0.397, ANCOVA; Mean Difference (Net) = -2.76, 95% CI 2-sided [-9.1631 to 3.6504], Standard Error of Mean 3.244
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #2 group based on the change from baseline at Day 14; Test type: Superiority; p = 0.804, ANCOVA; Mean Difference (Net) = 0.81, 95% CI 2-sided [-5.6006 to 7.2129], Standard Error of Mean 3.244
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #3 group based on the change from baseline at Day 14; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Net) = -9.32, 95% CI 2-sided [-15.7231 to -2.9096], Standard Error of Mean 3.244
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; Interpretation of between-treatment comparison between Wounded Uncovered group vs Product #4 group based on the change from baseline at Day 14; Test type: Superiority; p = 0.985, ANCOVA; Mean Difference (Net) = 0.06, 95% CI 2-sided [-6.3452 to 6.4683], Standard Error of Mean 3.244

37. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level- Baseline (Day 0)
Description: Quantification of oxy- and deoxy-hemoglobin at the wound area was achieved from apparent absorption spectrum acquired from diffuse reflectance spectroscopy (DRS) at the site. Absorption spectra of fully oxygenated and deoxygenated hemoglobin molecules were employed to quantify the contribution of each molecule to the total apparent absorption of the wounded skin in the spectral range of 560 nm -- 700 nm. The numbers of oxyhemoglobin are in arbitrary unit and higher values describe higher erythema levels.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 27 | 30 | 30 | 30 | 31 | 29
Arbitrary Unit | 0.82 (0.143) | 0.97 (0.189) | 0.96 (0.143) | 1.00 (0.198) | 0.99 (0.171) | 0.98 (0.179)

38. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 1
Description: as for outcome 37
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 25 | 26 | 26 | 27 | 27 | 27
Arbitrary Unit | 0.83 (0.127) | 1.20 (0.170) | 1.15 (0.181) | 1.12 (0.197) | 1.15 (0.178) | 1.22 (0.186)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.348, ANCOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.1290 to 0.0458], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 29, analysis 2]; Test type: Superiority; p = 0.019, ANCOVA; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.1904 to -0.0178], Standard Error of Mean 0.044
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 29, analysis 3]; Test type: Superiority; p = 0.183, ANCOVA; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.1437 to 0.0278], Standard Error of Mean 0.043
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 29, analysis 4]; Test type: Superiority; p = 0.736, ANCOVA; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.0725 to 0.1023], Standard Error of Mean 0.044

39. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 2
Description: as for outcome 37
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 26 | 27 | 27 | 27 | 27 | 27
Arbitrary Unit | 0.85 (0.100) | 1.21 (0.166) | 1.16 (0.181) | 1.07 (0.188) | 1.18 (0.218) | 1.37 (0.212)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 30, analysis 1]; Test type: Superiority; p = 0.516, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.1360 to 0.0687], Standard Error of Mean 0.052
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 30, analysis 2]; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.2459 to -0.0412], Standard Error of Mean 0.052
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 30, analysis 3]; Test type: Superiority; p = 0.671, ANCOVA; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.1235 to 0.0798], Standard Error of Mean 0.051
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 30, analysis 4]; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Net) = 0.15, 95% CI 2-sided [0.0504 to 0.2578], Standard Error of Mean 0.052

40. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 3
Description: as for outcome 37
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 14 | 17 | 16 | 16 | 17 | 15
Arbitrary Unit | 0.81 (0.156) | 1.16 (0.211) | 1.08 (0.121) | 1.06 (0.174) | 1.16 (0.160) | 1.33 (0.252)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.292, ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.1896 to 0.0579], Standard Error of Mean 0.062
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 31, analysis 2]; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.2773 to -0.0297], Standard Error of Mean 0.062
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 31, analysis 3]; Test type: Superiority; p = 0.538, ANCOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.1622 to 0.0853], Standard Error of Mean 0.062
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 31, analysis 4]; Test type: Superiority; p = 0.061, ANCOVA; Mean Difference (Net) = .012, 95% CI 2-sided [-0.0059 to 0.2515], Standard Error of Mean 0.065

41. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 4
Description: as for outcome 37
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 31 | 33 | 34 | 34 | 33 | 34
Arbitrary Unit | 0.81 (0.138) | 1.20 (0.166) | 0.99 (0.217) | 0.99 (0.205) | 1.14 (0.386) | 1.28 (0.252)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 32, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.3265 to -0.0895], Standard Error of Mean 0.060
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 32, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.3614 to -0.1243], Standard Error of Mean 0.060
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 32, analysis 3]; Test type: Superiority; p = 0.236, ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.1899 to 0.0471], Standard Error of Mean 0.060
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 32, analysis 4]; Test type: Superiority; p = 0.627, ANCOVA; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.0902 to 0.1492], Standard Error of Mean 0.061

42. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 5
Description: as for outcome 37
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24 | 23
Arbitrary Unit | 0.81 (0.159) | 1.14 (0.208) | 0.90 (0.146) | 0.96 (0.178) | 1.00 (0.207) | 1.26 (0.336)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.3331 to -0.1305], Standard Error of Mean 0.051
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 33, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.3091 to -0.1092], Standard Error of Mean 0.050
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 33, analysis 3]; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.2439 to -0.0457], Standard Error of Mean 0.050
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 33, analysis 4]; Test type: Superiority; p = 0.020, ANCOVA; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.0197 to 0.2252], Standard Error of Mean 0.052

43. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 6
Description: as for outcome 37
Time Frame: Day 6
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 30 | 30 | 28 | 29 | 29 | 29
Arbitrary Unit | 0.80 (0.124) | 1.20 (0.230) | 0.88 (0.146) | 0.95 (0.148) | 0.98 (0.159) | 1.23 (0.326)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.4019 to -0.2044], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 34, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.3655 to -0.1679], Standard Error of Mean 0.050
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 34, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.3338 to -0.1377], Standard Error of Mean 0.050
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 34, analysis 4]; Test type: Superiority; p = 0.646, ANCOVA; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.0767 to 0.1231], Standard Error of Mean 0.050

44. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 7
Description: as for outcome 37
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 32 | 33 | 33 | 33 | 33 | 33
Arbitrary Unit | 0.78 (0.111) | 1.02 (0.191) | 0.88 (0.164) | 0.89 (0.151) | 0.88 (0.141) | 1.03 (0.279)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 35, analysis 1]; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.2254 to -0.0384], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 35, analysis 2]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.2444 to -0.0574], Standard Error of Mean 0.047
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 35, analysis 3]; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.2541 to -0.0682], Standard Error of Mean 0.047
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 35, analysis 4]; Test type: Superiority; p = 0.911, ANCOVA; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.0891 to 0.0998], Standard Error of Mean 0.048

45. Secondary Outcome: Redness: Wound Area Oxyhemoglobin Level - Day 14
Description: as for outcome 37
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: Arbitrary Unit
Arm/Group | Intact Uncovered Skin | Wounded Uncovered Skin | Product #1 | Product #2 | Product #3 | Product #4
Number analyzed (Participants) | 29 | 30 | 28 | 29 | 29 | 29
Arbitrary Unit | 0.79 (0.120) | 0.90 (0.147) | 0.89 (0.146) | 0.85 (0.125) | 0.84 (0.112) | 0.92 (0.115)
Statistical Analysis 1: Comparison: Wounded Uncovered Skin vs Product #1; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.937, ANCOVA; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.0818 to 0.0755], Standard Error of Mean 0.040
Statistical Analysis 2: Comparison: Wounded Uncovered Skin vs Product #2; [analysis description as in outcome 36, analysis 2]; Test type: Superiority; p = 0.026, ANCOVA; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.1663 to -0.0108], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Wounded Uncovered Skin vs Product #3; [analysis description as in outcome 36, analysis 3]; Test type: Superiority; p = 0.045, ANCOVA; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.1562 to -0.0017], Standard Error of Mean 0.039
Statistical Analysis 4: Comparison: Wounded Uncovered Skin vs Product #4; [analysis description as in outcome 36, analysis 4]; Test type: Superiority; p = 0.956, ANCOVA; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.0799 to 0.0755], Standard Error of Mean 0.039

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time the informed consent was obtained through the subject's last study procedure/visit. Serious adverse events were collected through and including 30 calendar days after administration of the subject's last dose or exposure to IP.
Arm/Group | All Randomized Subjects
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03365934/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03365934/SAP_001.pdf